CLINICAL TRIAL: NCT06438900
Title: Fighting Western-diet Derived AGEs to Mitigate Muscle Wasting in Sarcobesity:Observational Study on the Relationship Between AGE Levels and Sarcobesity in an Adult Population Affected by Obesity and Type 2 Diabetes Mellitus
Brief Title: Investigating the Link Between Advanced Glycation End Products (AGEs) and Muscle Wasting in Sarcobesity
Acronym: Westernage
Status: Recruiting | Type: Observational
Sponsor: Azienda Ospedaliero Universitaria Maggiore della Carita (Other)
Responsible Party: Principal Investigator, Flavia Prodam, Professor, Azienda Ospedaliero Universitaria Maggiore della Carita
Other Study IDs: CE049/2024
Record Dates: First submitted 2024-05-14; First posted 2024-06-03 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Sarcopenia; Obesity
Keywords: Advanced glycation end products; Sarcobesity; Obesity; Sarcopenic
MeSH Terms: conditions — Sarcopenia; Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study aims to explore whether a high level of AGEs (Advanced Glycation end products) derived from the diet may mediate diet-related muscle loss in Western-type diet, influencing the onset and progression of sarcopenia, predisposing to earlier and more severe metabolic consequences, including type 2 diabetes (T2D).

The primary objective of the study is to investigate how the accumulation of AGEs is correlated with muscle loss in adult patients with obesity and type 2 diabetes or lipodystrophy in order to identify possible targets to mitigate the metabolic alterations caused by the Western diet (WD). Specifically, circulating AGEs levels on the skin will be evaluated and correlated with the stage of sarcopenia in a group of patients with obesity and a T2D diagnosis. Furthermore, the relationship between disease duration and AGE levels will be assessed.

A secondary objective will be to analyze the clinical data obtained to identify metabolites and metabolic pathways responsible for the phenotype induced by the WD.

The ultimate aim of the study is therefore to verify whether high levels of AGEs are correlated with an early and/or more pronounced onset of sarcopenia, concurrently with an increase in inflammation and oxidative stress.

DETAILED DESCRIPTION:
The study in question is of a cross-sectional observational type. The reference population is defined by patients with obesity and a diagnosis of T2D within 15 years of entry into the study or patients with concomitant type 2 diabetes and lipodystrophy syndrome. This population was chosen because they are at high risk of sarcopenia.

Lipodystrophy includes a heterogeneous spectrum of genetic and acquired diseases characterized by loss of subcutaneous adipose tissue, ectopic fat accumulation, insulin resistance, metabolic and cardiovascular diseases, premature aging, sarcopenia, muscle pain, high-grade inflammation, epigenetic dysregulation, and mitochondrial dysfunction. Therefore, patients with T2D and lipodystrophy are highly inflamed as they generally present with a more severe T2D phenotype, presumed sarcopenic, and with a high rate of endogenous AGE production. Patients with concurrent lipodystrophy and T2D will be recruited as sarcopenic and obese subjects, representing an excellent strategy for comparison with diabetic individuals without lipodystrophy.

SUBJECTS AND METHODS A total of 195 consecutive subjects will be enrolled in the study from the Endocrinology Unit of the University of Eastern Piedmont between April 2024 and April 2026, who meet the inclusion criteria.

Study duration:

The study will last for two years corresponding to the enrollment period given the cross-sectional nature of the study.

Statistical Analysis

Descriptive statistics will be used to summarize sociodemographic, anthropometric, clinical, and lifestyle-related information collected. Categorical variables will be summarized using absolute frequencies and percentages, while numerical variables will be summarized using mean and standard deviation or median and interquartile range if not normally distributed according to the Shapiro-Wilk test and after observation of Q-Q plots (quantile-quantile plot).

The Pearson correlation coefficient or the corresponding non-parametric Spearman rank correlation coefficient and confidence intervals will be initially calculated to assess the correlation between the levels of individual AGEs and skeletal muscle mass (SMM), handgrip strength (HGS), parameters of body composition, and functional parameters of skeletal muscle. Subsequently, linear regression models will be used to evaluate the relationship between AGEs and sarcopenia-defining indices adjusted for age, sex, duration of diabetes, and other potential confounding factors such as inflammation, adherence to the Western diet, and levels of physical activity. The LASSO method will be used for variable selection in multivariable regression models.

Univariable and multivariable Poisson regression models with robust variance will be used to estimate relative prevalence risks for the association between AGEs and patient characteristics with sarcopenia presence and the corresponding confidence intervals.

An integration of clinical data, biochemical data, AGE levels, and patient omic signatures will be performed to develop a multifactorial diagnostic model using multivariate statistical analysis (e.g., factor analysis, principal component analysis, cluster analysis, discriminant analysis, partial least squares analysis, logistic regression) and data-driven approaches. Machine learning algorithms will be applied to prioritize and weigh risk factors. These analyses will be conducted with internal statistical consultation already utilized by the group.

Expected Results

With this study, the investigators expect to obtain further information and correlations between nutritional assessment and its impact on inflammation, sarcopenia definition, and progression, obesity, and T2D, based on body measurements and clinical parameters. Through biochemical, hormonal, and metabolomic analyses conducted on biological samples, te investigators expect to identify possible markers related to the presence of AGEs. In conclusion, the primary expected outcome would be to identify a positive correlation between AGE accumulation in at least one compartment (skin, plasma, urine) and the severity of sarcopenia, thus obtaining a rapid and non-invasive method to identify individuals at high risk of developing muscle wasting (MW) and identify correlations between AGE levels and other metabolic characteristics, even in lipodystrophic pathology.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes.
* Adults.
* BMI compatible with obesity and a diagnosis of type 2 diabetes under good metabolic control (HbA1c < 7.5%) within 15 years of entry into the study or diagnosis of lipodystrophy (included in the European Consortium of Lipodystrophies (ECLip) Registry (eclip-web.org))

Exclusion Criteria:

* Age under 18 years.
* Secondary obesity or genetic diseases (Prader-Willi Syndrome, Down Syndrome); metabolic and endocrine disorders (Cushing's syndrome, hypothyroidism).
* Subjects with: Inflammatory Bowel Disease (IBD), cancer.
* Confirmed or planned pregnancy during the study participation months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Given a type I error rate (α) of 0.05 and a power of 80%, 195 subjects will be needed to observe a significant correlation between AGE levels and sarcobesity indices of at least 0.2. Considering the low prevalence of lipodystrophy and a recruitment duration of one year, approximately 35 subjects with this condition are expected to be included. The remaining 160 subjects will have diabetes and obesity. Furthermore, considering that the duration of diabetes may influence AGE levels and sarcobesity, both subjects with long-standing diabetes (80 patients) and those with less than one year of diagnosis (80 patients) will be selected, which can be considered comparable to subjects in pre-diabetes.
Sampling Method: Probability Sample
Enrollment: 195 (Estimated)
Dates: Start 2024-06-15 (Actual); Primary Completion 2026-05-15 (Estimated); Study Completion 2026-05-15 (Estimated)

PRIMARY OUTCOMES:
Skeletal mass functionality for sarcopenia definition | evaluation of sarcopenia state through study completion, an average of 1 year
  Functional parameters of skeletal muscle defined by muscle strength measured through hand grip strength (HGS) The test requires the patient to tighten the handle the dynamometer with the maximum possible force, then maintaining the contraction for at least 5 seconds; you should repeat the test on the other hand (it is normal that the dominant expresses a higher force) and possibly repeat the test 2-3 times, with a break between different attempts, then going to calculate the average oh the kg moved with the dynamometer
Skeletall mass fuctionality for sarcopenia definition | evaluation of sarcopenia state through study completion, an average of 1 year
  Functional parameters of skeletal muscle defined by the chair test: five-times sit-to-stand test; time duration 30-second chair stand test. You measure by considering the ability in seconds to get up and sit down from the chair properly
Skeletall mass calculation for sarcopenia definition | evaluation of sarcopenia state through study completion, an average of 1 year
  The percentage of skeletal muscle mass relative to body mass will be considered.
  Skeletal mass will be calculated as follows:
  SM(Kg)=[(h^2/(BIA resistance)0.401)+(gender3.825)+(age*0.071)]+5.102 Where h indicates height measured in cm, gender is a dichotomous variable taking a value of 1 for males and 0 for females, and age is measured in years.
  From this measurement, the percentage of skeletal muscle mass (%SMM) will be calculated:
  %SMM=(SM (Kg))/(Body mass (Kg))*100
Number of participants with sarcopenia | evaluation of sarcopenia state through study completion, an average of 1 year
  According to consensus statement of European Society for Clinical Nutrition and Metabolism (ESPEN) and dell' European Association for the Study of Obesity (EASO) guidelines, individuals with altered skeletal muscle functionality parameters (HGS < 16 kg for females and < 27 kg for males or chair test >15 seconds for both males and females [27]), altered %BF(body fat) (≥ 25% for males and ≥35% for females [28]), and altered %SMM (<35.6% (≤28.7% severe sarcopenia) for males, <28.4% (≤23% severe sarcopenia) for females) will be defined as sarcopenic.
Advanced glycation end products quantification | evaluation of AGEs through study completion, an average of 1 year
  AGE levels will be measured using skin fluorescence, using the "AGE reader mu" device (range from 1.3 to 5 level of AGEs respect to the patient's age).
Endogenous and exogenous AGEs plasma quantification | evaluation of AGEs through study completion, an average of 1 year
  AGEs will also be assessed at the plasma level in free form (ELISA, fluorescence assay) or bound to hemoglobin (HbA1c clinical practice test), both measured in pg/mL

SECONDARY OUTCOMES:
With questionnaires assessment of socio-demographic characteristics | evaluation of socio-demographic characteristics through study completion, an average of 1 year
  Gender, date of birth, date of diabetes diagnosis (for diabetic subjects) are assessed through questionnaires and medical record
Anthropometric measurements | evaluation of weight and body composition through study completion, an average of 1 year
  weight is assessed in Kg with the use of the bioimpedance balance
Anthropometric measurements | evaluation of height through study completion, an average of 1 year
  the height is measured in cm through a wall altimeter
Anthropometric measurements | evaluation of BMI (body mass index) through study completion, an average of 1 year
  the BMI (body mass index) is calculated by making the ratio of the weight to the square of the height
Anthropometric measurements | evaluation of circumferences through study completion, an average of 1 year
  waist, hip, arm, and calf circumference are measured using an anelastic meter
Dietary Inflammatory Index (DII) | evaluation of DII through study completion, an average of 1 year
  Calculated using Alternative Healthy Eating Index-2010 (AHEI-2010) derived from basal metabolism assessment through fasting morning indirect calorimetry.
Adherence level to the Western diet with European Prospective Investigation into Cancer and Nutrition (EPIC) questionnaires | evaluation of DII through study completion, an average of 1 year
  Assessed with the use of questionnaire. EPIC is used for the bromatology evaluation of the diet, so there aren't scales but only indication about the macro and micronutrient composition. This is a qualitative questionnaires and not quantitative.
Adherence level to the Western diet with 24h recall questionnaires | evaluation of DII through study completion, an average of 1 year
  Assessed with the use of questionnaires. 24h recall questionnaire is used for the bromatology evaluation of the diet, so there aren't scales but only indication about the macro and micronutrient composition. This is a qualitative questionnaires and not quantitative.
Level of physical activity, related to sarcopenia,using a questionnaire | evaluation of METs through study completion, an average of 1 year
  Physical activity is assessed using the International Physical Activity Questionnaire (IPAQ), which provides results in Metabolic Equivalent of Tasks (METs). The questions refer to activities over the past 7 days, including work, transportation, and leisure time.
  Moderate physical activity: Requires moderate effort and a slightly higher breathing rate than normal. One can speak but not sing during this activity.
  Intense physical activity: Requires significant effort and a much higher breathing rate, causing sweating and making it difficult to talk.
  The METs scale is as follows:
  Less than 700 METs: Inactive 700 to 2519 METs: Sufficiently active More than 2520 METs: Active

CONTACTS AND LOCATIONS:
Overall Officials: Flavia Prodam, MD PhD, Principal Investigator — AOU Maggiore della Carità di Novara
Locations (1):
- SCDU Endocrinology, AOU Ospedale Maggiore della Carità, Novara, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Frontera WR, Ochala J. Skeletal muscle: a brief review of structure and function. Calcif Tissue Int. 2015 Mar;96(3):183-95. doi: 10.1007/s00223-014-9915-y. Epub 2014 Oct 8. PMID 25294644
- [Background] Merz KE, Thurmond DC. Role of Skeletal Muscle in Insulin Resistance and Glucose Uptake. Compr Physiol. 2020 Jul 8;10(3):785-809. doi: 10.1002/cphy.c190029. PMID 32940941
- [Background] Bonaldo P, Sandri M. Cellular and molecular mechanisms of muscle atrophy. Dis Model Mech. 2013 Jan;6(1):25-39. doi: 10.1242/dmm.010389. PMID 23268536
- [Background] Cohen S, Nathan JA, Goldberg AL. Muscle wasting in disease: molecular mechanisms and promising therapies. Nat Rev Drug Discov. 2015 Jan;14(1):58-74. doi: 10.1038/nrd4467. PMID 25549588
- [Background] Dutt V, Gupta S, Dabur R, Injeti E, Mittal A. Skeletal muscle atrophy: Potential therapeutic agents and their mechanisms of action. Pharmacol Res. 2015 Sep;99:86-100. doi: 10.1016/j.phrs.2015.05.010. Epub 2015 Jun 2. PMID 26048279
- [Background] Lecker SH, Jagoe RT, Gilbert A, Gomes M, Baracos V, Bailey J, Price SR, Mitch WE, Goldberg AL. Multiple types of skeletal muscle atrophy involve a common program of changes in gene expression. FASEB J. 2004 Jan;18(1):39-51. doi: 10.1096/fj.03-0610com. PMID 14718385
- [Background] Hosseini Z, Whiting SJ, Vatanparast H. Current evidence on the association of the metabolic syndrome and dietary patterns in a global perspective. Nutr Res Rev. 2016 Dec;29(2):152-162. doi: 10.1017/S095442241600007X. PMID 27955720
- [Background] Tsilingiris D, Tzeravini E, Koliaki C, Dalamaga M, Kokkinos A. The Role of Mitochondrial Adaptation and Metabolic Flexibility in the Pathophysiology of Obesity and Insulin Resistance: an Updated Overview. Curr Obes Rep. 2021 Sep;10(3):191-213. doi: 10.1007/s13679-021-00434-0. Epub 2021 Apr 10. PMID 33840072
- [Background] Peppa M, Mavroeidi I. Experimental Animal Studies Support the Role of Dietary Advanced Glycation End Products in Health and Disease. Nutrients. 2021 Sep 29;13(10):3467. doi: 10.3390/nu13103467. PMID 34684468
- [Background] Muthyalaiah YS, Jonnalagadda B, John CM, Arockiasamy S. Impact of Advanced Glycation End products (AGEs) and its receptor (RAGE) on cancer metabolic signaling pathways and its progression. Glycoconj J. 2021 Dec;38(6):717-734. doi: 10.1007/s10719-021-10031-x. Epub 2022 Jan 22. PMID 35064413
- [Background] Mori H, Kuroda A, Ishizu M, Ohishi M, Takashi Y, Otsuka Y, Taniguchi S, Tamaki M, Kurahashi K, Yoshida S, Endo I, Aihara KI, Funaki M, Akehi Y, Matsuhisa M. Association of accumulated advanced glycation end-products with a high prevalence of sarcopenia and dynapenia in patients with type 2 diabetes. J Diabetes Investig. 2019 Sep;10(5):1332-1340. doi: 10.1111/jdi.13014. Epub 2019 Feb 19. PMID 30677242
- [Background] Waqas K, Chen J, Trajanoska K, Ikram MA, Uitterlinden AG, Rivadeneira F, Zillikens MC. Skin Autofluorescence, a Noninvasive Biomarker for Advanced Glycation End-products, Is Associated With Sarcopenia. J Clin Endocrinol Metab. 2022 Jan 18;107(2):e793-e803. doi: 10.1210/clinem/dgab632. PMID 34453164
- [Background] Chiu CY, Yang RS, Sheu ML, Chan DC, Yang TH, Tsai KS, Chiang CK, Liu SH. Advanced glycation end-products induce skeletal muscle atrophy and dysfunction in diabetic mice via a RAGE-mediated, AMPK-down-regulated, Akt pathway. J Pathol. 2016 Feb;238(3):470-82. doi: 10.1002/path.4674. Epub 2015 Dec 31. PMID 26586640
- [Background] Chiappalupi S, Sorci G, Vukasinovic A, Salvadori L, Sagheddu R, Coletti D, Renga G, Romani L, Donato R, Riuzzi F. Targeting RAGE prevents muscle wasting and prolongs survival in cancer cachexia. J Cachexia Sarcopenia Muscle. 2020 Aug;11(4):929-946. doi: 10.1002/jcsm.12561. Epub 2020 Mar 11. PMID 32159297
- [Background] Egawa T, Tsuda S, Goto A, Ohno Y, Yokoyama S, Goto K, Hayashi T. Potential involvement of dietary advanced glycation end products in impairment of skeletal muscle growth and muscle contractile function in mice. Br J Nutr. 2017 Jan;117(1):21-29. doi: 10.1017/S0007114516004591. Epub 2017 Jan 17. PMID 28093090
- [Background] Mastrocola R, Nigro D, Chiazza F, Medana C, Dal Bello F, Boccuzzi G, Collino M, Aragno M. Fructose-derived advanced glycation end-products drive lipogenesis and skeletal muscle reprogramming via SREBP-1c dysregulation in mice. Free Radic Biol Med. 2016 Feb;91:224-35. doi: 10.1016/j.freeradbiomed.2015.12.022. Epub 2015 Dec 22. PMID 26721591
- [Background] Clayton ZS, Gioscia-Ryan RA, Justice JN, Lubieniecki KL, Hutton DA, Rossman MJ, Zigler MC, Seals DR. Lifelong physical activity attenuates age- and Western-style diet-related declines in physical function and adverse changes in skeletal muscle mass and inflammation. Exp Gerontol. 2022 Jan;157:111632. doi: 10.1016/j.exger.2021.111632. Epub 2021 Nov 22. PMID 34822971
- [Background] Roseno SL, Davis PR, Bollinger LM, Powell JJ, Witczak CA, Brault JJ. Short-term, high-fat diet accelerates disuse atrophy and protein degradation in a muscle-specific manner in mice. Nutr Metab (Lond). 2015 Nov 4;12:39. doi: 10.1186/s12986-015-0037-y. eCollection 2015. PMID 26539241
- [Background] M V, Wang K. Dietary natural products as a potential inhibitor towards advanced glycation end products and hyperglycemic complications: A phytotherapy approaches. Biomed Pharmacother. 2021 Dec;144:112336. doi: 10.1016/j.biopha.2021.112336. Epub 2021 Oct 19. PMID 34678719
- [Background] Garvey WT. New Horizons. A New Paradigm for Treating to Target with Second-Generation Obesity Medications. J Clin Endocrinol Metab. 2022 Mar 24;107(4):e1339-e1347. doi: 10.1210/clinem/dgab848. PMID 34865050
- [Background] Donini LM, Busetto L, Bischoff SC, Cederholm T, Ballesteros-Pomar MD, Batsis JA, Bauer JM, Boirie Y, Cruz-Jentoft AJ, Dicker D, Frara S, Fruhbeck G, Genton L, Gepner Y, Giustina A, Gonzalez MC, Han HS, Heymsfield SB, Higashiguchi T, Laviano A, Lenzi A, Nyulasi I, Parrinello E, Poggiogalle E, Prado CM, Salvador J, Rolland Y, Santini F, Serlie MJ, Shi H, Sieber CC, Siervo M, Vettor R, Villareal DT, Volkert D, Yu J, Zamboni M, Barazzoni R. Definition and Diagnostic Criteria for Sarcopenic Obesity: ESPEN and EASO Consensus Statement. Obes Facts. 2022;15(3):321-335. doi: 10.1159/000521241. Epub 2022 Feb 23. PMID 35196654
- [Background] Donini LM, Poggiogalle E, Del Balzo V, Lubrano C, Faliva M, Opizzi A, Perna S, Pinto A, Rondanelli M. How to estimate fat mass in overweight and obese subjects. Int J Endocrinol. 2013;2013:285680. doi: 10.1155/2013/285680. Epub 2013 Apr 10. PMID 23662101
- [Background] De Rosa E, Santarpia L, Marra M, Sammarco R, Amato V, Onufrio M, De Simone G, Contaldo F, Pasanisi F. Preliminary evaluation of the prevalence of sarcopenia in obese patients from Southern Italy. Nutrition. 2015 Jan;31(1):79-83. doi: 10.1016/j.nut.2014.04.025. Epub 2014 May 10. PMID 25441590

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-04-15): https://cdn.clinicaltrials.gov/large-docs/00/NCT06438900/Prot_SAP_000.pdf